CLINICAL TRIAL: NCT03095989
Title: An Online Mindfulness Intervention for People With ALS and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Collaborators: ALS Association (Other); Milton S. Hershey Medical Center (Other); Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Francesco Pagnini, Post-Doctoral Fellow, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB14-3695
Record Dates: First submitted 2016-03-24; First posted 2017-03-30 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: mindfulness
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness (Experimental): Subjects in the intervention group will participate in an online mindfulness program developed in the first phase of the study, in addition to standard clinical care.
  Interventions: Behavioral: Mindfulness
- Waiting list (No Intervention): Participants from the control group will be placed on a waiting list and will receive the standard care, that they would receive if not in the study. They will be assessed according to the assessment schedule, exactly as subjects in the intervention group. After the last assessment (six months after recruitment), they will receive the option to enter the mindfulness program.

INTERVENTIONS:
Behavioral: Mindfulness — The structure of the protocol incorporates key features of Langer's mindfulness theory. Many of the tasks and exercises have demonstrated increased mindfulness in the general population and have been modified to incorporate ALS-specific exercises that make sense from patients and caregivers' points of view. The intervention provides easily understood multimedia (video and written) presentations of the framework of mindfulness and the aims of the planned tasks. The general structure of the protocol mixes different mindfulness elements; for every week there is a specific topic examined in depth. These topics are: Attention to variability; Positive and negative events; Unpredictability; Sense Making; and Novelty seeking / novelty producing. The overall duration of the protocol is 5 weeks.
  Arms: Mindfulness

SUMMARY:
The psychological impact of ALS on both patients and caregivers is high and affects their quality of life (QOL). However, there is minimal research about psychological interventions to improve QOL in the ALS scientific literature.

Recent advances in clinical treatments aimed at improving the health of people with chronic disorders are based on the concept of mindfulness. Mindfulness can be defined as a flexible state of mind resulting from the simple act of actively noticing new things, as opposed to mindlessness, the human tendency to operate on" autopilot".

Preliminary data suggests that mindfulness may promote a better QOL for people with ALS and their caregivers. The investigators also found that a mindful attitude was associated with slower disease progression.

This project's goal is to develop an innovative, web-based online mindfulness training program and intervention, customized for people with ALS and their primary caregivers. It is an active learning intervention, with cognitive exercises and lectures that increase participants' mindfulness. The efficacy of this program for improving QOL, and for reducing anxiety and depression in people with ALS and their caregivers, will be tested with a randomized clinical trial. Assessments immediately post-treatment as well as 3 and 6 months after recruitment will be conducted, comparing subjects undergoing the mindfulness intervention to a control group.

DETAILED DESCRIPTION:
Quality of Life in people with ALS is not related to physical function, but is related to psychological, existential, and support factors. ALS caregivers demonstrate considerable burden and low QOL. It has been proposed by the investigators that it is time for the ALS field to develop "best practices" that use psychological intervention to improve QOL, reducing psychological distress in people with ALS and their caregivers. A disease that is as inexorably progressive and physically devastating as ALS also inevitably has an immense psychological impact on caregivers, both at the time of diagnosis and throughout the course of the disease. Yet, there is scant research on psychological interventions for ALS patients and caregivers.

Over 35 years of research demonstrate that mindfulness-based interventions comprise some of the most promising behavioral treatments in QOL improvement for people with chronic disorders.This work is based on socio-cognitive aspects of mindfulness, conceptualized as having a flexible state of mind that incorporates active engagement in the present and being sensitive to context and perspective. In over 35 years of research it has been shown that a higher state of mindfulness correlates with an improved QOL. In addition, mindfulness may lead to an improvement in some physiological as well as psychological measures. The literature on mindfulness in other disorders, combined with preliminary data on mindfulness in ALS patients and their caregivers, provides a strong evidence-based platform for proposing a careful study of the effects of mindfulness on psychological and physiological measures of ALS patients and their caregivers. The investigators conducted an exploratory investigation on a large sample (100+) of people with ALS about the influence of mindfulness on QOL and the course of the disease. The investigators found that mindfulness predicted positive QOL and psychological well-being, reducing anxiety and depression. That was quite expected. However, another finding was that mindfulness positively influenced the changes in physical symptoms: subjects with higher mindfulness experienced a slower progression of the disease, as measured by the self- administered ALS Functional Rating Scale (SA-ALSFRS). Furthermore, mindfulness was a significant predictor of positive QOL and psychological well-being in ALS caregivers, with a protective effect against anxiety and depression.

Fifty (50) participants with ALS, together with each subject's primary caregiver (i.e., an expected overall sample of 100 subjects), will be directly recruited from the Hershey Medical Center ALS Clinic at Penn State University. Participants will sign IRS-approved informed consent documents. Both patients and caregivers may be recruited even if a component of the dyad (patient-caregiver) opts not to join the study (i.e. patients and caregivers alone may be recruited). ALS patient-caregiver couples will be considered as a single subject for randomisation purposes (meaning that both the patient and the caregiver are randomly allocated to the same group). Subjects will be randomized into two groups (employing true randomization from atmospheric noise, www.random.org): an intervention group and a control group. Subjects in the intervention group will participate in the online mindfulness program, in addition to standard clinical care.

The intervention for each patient-caregiver pair will commence immediately after recruitment, on a rolling basis. Participants from the control group will be placed on a waiting list and will receive the standard care that they would receive if not in the study. Participants from both groups will be assessed 4 times: at recruitment (T1, baseline); after completing the intervention, or 5 weeks after recruitment for the control group (T2, post- treatment); three months after recruitment (T3); six months after recruitment (T4).

The primary outcome measure will be QOL (assessed with the ALS-Specific Quality of Life-Revised instrument, the ALSSQOL-R) in ALS subjects. Secondary outcomes from ALS subjects will be: depression and anxiety (assessed with the Hospital Anxiety and Depression Scale), attained mindfulness level (assessed with the Langer Mindfulness Scale) functional, cognitive and respiratory variables, assessed respectively with the Self-Administered ALS Functional Rating Scale-Revised, the Edinburgh Cognitive Assessment and Forced Vital Capacity. Caregivers outcomes, considered as secondary outcomes, will be QOL (assessed with the Short Form-36), depression and anxiety (assessed with the Hospital Anxiety and Depression Scale), care burden (assessed with the Zarit Burden Inventory) and mindfulness (assessed with the Langer Mindfulness Scale). A sub-sample of the subjects from the intervention group may be invited to a semi-structured interview about the experience with the treatment.

After the last assessment, subjects in the control group will have the option to enter the mindfulness program. All the subjects will have the option to continue to use the program after the 5-week intervention.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for ALS Subjects:

* Definite, probable, probable laboratory-supported, or possible ALS by revised El-Escorial criteria (Brooks, Miller, Swash, & Munsat, 2000).
* Must have the physical ability, with or without adaptive devices, to use a computer and access the Internet.
* A forced vital capacity of 50% or greater than the predicted value, measured within 30 days of enrollment. If impaired bulbar function compromises accurate pulmonary function testing as determined by the study neurologist, then a forced vital capacity as low as 40% of predicted is permitted. If taken, stable doses of anti-anxiety or antidepressant medications for 30 days before study entry, and during the study from the T1 to the T2 time point.

Inclusion Criteria for Caregivers:

* Must have the physical ability to use a computer and access the Internet.

Exclusion Criteria:

Exclusion Criteria for ALS Subjects:

* Scores on the Edinburgh Cognitive Assessment (ECAS) within 90 days of study entry, that meet criteria for mild frontotemporal dysfunction (either cognitive or behavioral)
* Significant cognitive impairment or significant uncontrolled psychiatric disease (for example, schizophrenia, bipolar disorder), in the opinion of the study neurologist.
* Unsuitable for the study as determined by the study neurologist.
* Regular meditation or participation in a mindfulness program in past 6 months.

Exclusion Criteria for Caregivers:

* Unwillingness to participate in the study
* Unsuitable for the study as determined by the clinical staff. For example, the clinical staff may consider inappropriate a caregiver who showed no real interest toward the care process or showed signs of severe mental health problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 4-6 weeks after recruitment
  ALS-Specific Quality of Life-Revised (ALSSQoL-R; Simmons et al., 2006)

SECONDARY OUTCOMES:
Depression and anxiety | Baseline (T1); one month after recruitment (T2); three months after recruitment (T3); six months after recruitment (T4)
  Hospital Anxiety and Depression Scale (HADS; Zigmond & Snaith, 1983)
Quality of Life | Baseline (T1); three months after recruitment (T3); six months after recruitment (T4)
  ALS-Specific Quality of Life-Revised (ALSSQoL-R; Simmons et al., 2006)
The patient's perception of physical impairment | Baseline (T1); one month after recruitment (T2); three months after recruitment (T3); six months after recruitment (T4)
  the Self-Administered ALS Functional Rating Scale-Revised (SA-ALSFRS; Montes et al., 2006)
Physician-assessed physical impairment | Baseline (T1); three months after recruitment (T3); six months after recruitment (T4)Baseline (T1); 4-6 weeks after recruitment (T2); three months after recruitment (T3); six months after recruitment (T4)
  ALS Functional Rating Scale-Revised (ALSFRS-R; Cedarbaum, et al., 1999)
Vital capacity (VC) | Baseline (T1); three months after recruitment (T3); six months after recruitment (T4)Baseline (T1); 4-6 weeks after recruitment (T2); three months after recruitment (T3); six months after recruitment (T4)
  Spirometer
Cognitive and behavioral function | Baseline (T1); three months after recruitment (T3); six months after recruitment (T4)Baseline (T1); 4-6 weeks after recruitment (T2); three months after recruitment (T3); six months after recruitment (T4)
  Edinburgh Cognitive Assessment (Abrahams et al., 2014)
Caregiver burden (caregivers only) | Baseline (T1); one month after recruitment (T2); three months after recruitment (T3); six months after recruitment (T4)
  Zarit Burden Inventory (ZBI; Zarit, Reever, & Bach-Peterson, 1980)

OTHER OUTCOMES:
Mindfulness | Baseline (T1); 4-6 weeks after recruitment (T2); three months after recruitment (T3); six months after recruitment (T4)
  Langer Mindfulness Scale (LMS; Pirson, Langer et al., 2012)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Langer, PhD, Principal Investigator — Professor of Psychology
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pagnini F, Phillips D, Bosma CM, Reece A, Langer E. Mindfulness as a Protective Factor for the Burden of Caregivers of Amyotrophic Lateral Sclerosis Patients. J Clin Psychol. 2016 Jan;72(1):101-11. doi: 10.1002/jclp.22235. Epub 2015 Oct 20. PMID 26485696
- [Background] Pagnini F, Phillips D, Bosma CM, Reece A, Langer E. Mindfulness, physical impairment and psychological well-being in people with amyotrophic lateral sclerosis. Psychol Health. 2015;30(5):503-17. doi: 10.1080/08870446.2014.982652. Epub 2014 Nov 26. PMID 25361013